CLINICAL TRIAL: NCT06316479
Title: A Prospective, Multi-Centre, Single-Arm First-In-Man Study to Evaluate the Safety and Performance of PTMC Dermal Filler for the Correction of Moderate to Severe Nasolabial Folds
Brief Title: Safety and Performance of PTMC Dermal Filler
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Aqpha Medical B.V. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CI-001-23
Record Dates: First submitted 2024-03-12; First posted 2024-03-18 (Actual); Last update posted 2024-03-18 (Actual); Status verified 2024-03

CONDITIONS: Moderate to Severe Nasolabial Fold

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment group (Experimental): All participants will receive PTMC Dermal Filler.
  Interventions: Device: PTMC Dermal Filler

INTERVENTIONS:
Device: PTMC Dermal Filler — A total of 120 subjects will receive treatment with PTMC Dermal Filler. The volume of filler injected will vary depending on the severity of the nasolabial fold. Injections will be administered by the investigator at the beginning of the study, with the injection technique, plane, and volume recorded. Touch-up treatments are permitted at the 1-month follow-up visit, if necessary.

SUMMARY:
The goal of this clinical trial is to assess the safety and performance of the PTMC Dermal filler for treating moderate to severe nasolabial folds in adult men and women.

The main questions it aims to answer are:

* Does the PTMC dermal filler maintain its performance for a minimum of 6 months?
* Is the treatment considered safe for participants?

Participants will:

* Before treatment, the investigator will assess your medical history, medication usage, and satisfaction with your wrinkles/folds.
* You'll receive one injection of the PTMC Dermal filler during your initial visit.
* For 30 days post-injection, you'll keep a diary to note any reactions like pain, redness, or swelling at the injection site.
* At the 1-month follow-up, you can request a 'touch-up' of the filler, extending your participation in the study.
* Participants will visit the clinic a total of 8 times, including the initial treatment and 7 follow-up visits, spanning up to 18 months.
* Each visit will last approximately 60-90 minutes. The visits will be conducted in person.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female ≥18 years and £67 old.
2. Two fully visible bilateral nasolabial folds each with a Wrinkle Severity Rating Scale (WSRS) score of 3 or 4 that may be corrected with an injectable dermal filler.
3. If female and of childbearing potential: a negative urine pregnancy test + agreement to use adequate contraception.
4. Ability to understand and comply with the study requirements.
5. Willingness and ability to provide written informed consent.
6. Agree to refrain from seeking other treatment of nasolabial folds during the study.
7. Over the counter (OTC) wrinkle products or prescription wrinkle treatments, if used, shall be continued throughout the study in similar manner as performed prior to participation.

Exclusion Criteria:

1. Wrinkle Severity Rating Scale (WSRS) score of ≤ 2 on the right or left nasolabial fold.
2. Women who are pregnant or lactating or planning to become pregnant during the study.
3. Evidence of scar-related disease or delayed healing activity within the past 1 year.
4. History of keloid formation or hypertrophic scars.
5. Scars at the intended treatment sites.
6. Any infection or wound on the face.
7. Facial tattoo that may interfere with diagnosis.
8. Allergic history including anaphylaxis or multiple severe allergies to natural rubber latex or lidocaine.
9. Clinically significant organic disease including clinically significant cardiovascular, hepatic, pulmonary, neurologic, or renal disease or other medical condition, serious intercurrent illness, or extenuating circumstance that, in the opinion of the investigator preclude participation in the trial.
10. Aspirin, or nonsteroidal anti-inflammatory drugs within 1 week (7 days) prior to treatment.
11. Systemic (oral/injectable) corticosteroids or immunosuppressive medications within 30 days prior to treatment and topical steroids on the face within 14 days prior to trial start and throughout the study.
12. Concomitant anticoagulant therapy, antiplatelet therapy, biotherapy or history of bleeding disorders or connective tissue disorders.
13. Immunocompromised or immunosuppressed.
14. History of autoimmune diseases.
15. Anti-covid vaccination (RNA-based vaccines) within 2 weeks (14 days) prior to treatment.
16. Received any investigational product within 30 days prior to treatment.
17. Received prior dermabrasion, or botulinum toxins under the orbital rim (tear through) within 6 months (180 days) prior to entry into the study.
18. Received facelift within 2 years prior to treatment.
19. Previous tissue augmentation (bulking agents) for facial wrinkles and scars within 6 months at the mid-face.
20. Previous tissue augmentation with permanent implants.
21. Treatment of microdermabrasion or micro needling within the whole facial area within 3 months prior to treatment.
22. Laser treatment within the whole facial area within 6 months prior to treatment.

Ages: 18 Years to 67 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2024-08 (Estimated); Primary Completion 2024-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Nasolabial fold severity | 6 months after treatment
  The nasolabial fold severity is measured using the Wrinkles Severity Rating Scale (WSRS) by the investigator.

SECONDARY OUTCOMES:
Safety (Adverse events) | until 18 months after treatment
  Safety is assessed by the collection of adverse events (incidence and severity), and through subject assessment of injection site responses (ISRs) up to 4 weeks after treatment.
Nasolabial fold severity | 1, 3, 9, 12, and 18 months after treatment
  Mean change from baseline of the nasolabial fold severity measured using the WSRS by the investigator.
Responder rate | 1, 3, 6, 9, 12, and 18 months after treatment
  Number of subjects having at least 1-point improvement in the WSRS score compared to the baseline.
Overall aesthetic improvement (by the investigator) | 1, 3, 6, 9, 12, and 18 months after treatment
  Overall aesthetic improvement is assessed by the investigator using the Global Aesthetic Improvement Scale (GAIS).
Overall aesthetic improvement (by the subject) | 1, 3, 6, 9, 12, and 18 months after treatment
  Overall aesthetic improvement assessed by the subject using the Global Aesthetic Improvement Scale (GAIS).
Subject satisfaction | 1, 3, 6, 9, 12, and 18 months after treatment
  Subject satisfaction is measured using a FACE-Q questionnaire.

OTHER OUTCOMES:
Visual Analog Scale (VAS) for pain | After each injection and at the 2-weeks follow-up visit
  Evaluation of pain by the participant using Visual Analog Scale (VAS)
Treatment satisfaction | 1, 3, 6, 9, 12, and 18 months after treatment
  Treatment satisfaction evaluated by the subject using a questionnaire.
Ease of use | After injection of the device on day 0
  Ease of use of the device evaluated by the investigator using a questionnaire.